CLINICAL TRIAL: NCT00500851
Title: Evaluation of Two Methods of Jejunal Placement of Enteral Feeding Tubes in Critically Ill Patients: Endoscopic Versus Electromagnetic Method (CORTRAK™)
Brief Title: Evaluation of Jejunal Placement of Enteral Feeding Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Ulrike Holzinger, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 138/2007
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2009-02

CONDITIONS: Critical Illness; Tube Feeding
Keywords: critical illness; enteral nutrition; gastrointestinal intubation
MeSH Terms: conditions — Critical Illness | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): In case of meeting clinical criteria for jejunal feeding, tubes are placed using CORTRAK (electromagnetic imaging).
  Interventions: Device: Electromagnetic imaging for jejunal tube placement (CORTRAK)
- 2 (Active Comparator): Endoscopic placement of jejunal feeding tubes fulfilling clinical indication for jejunal feeding.
  Interventions: Device: Endoscopy

INTERVENTIONS:
Device: Electromagnetic imaging for jejunal tube placement (CORTRAK) — Jejunal feeding tubes are placed using electromagnetic imaging (CORTRAK)
  Other Names: CORTRAK
  Arms: 1
Device: Endoscopy — Endoscopic placement of jejunal feeding tubes
  Other Names: Endoscopy (Olympus); FREKA Trelumina
  Arms: 2

SUMMARY:
The purpose of this study is the evaluation of the success rate of jejunal tube placement comparing the endoscopic versus the electromagnetic method in a comparative ICU patient population. The investigators hypothesized that success rate of the electromagnetic jejunal tube placement will be lower than the success rate of the endoscopic method.

DETAILED DESCRIPTION:
Clinical studies have shown that up to 62,8% of patients receiving EN have gastrointestinal complications like high gastric residuals (≥200ml), vomiting, abdominal distension and regurgitation. These complications lead to interruptions of the EN, which result in a low caloric intake of the patient.

In order to avoid at least some of these complications the ACCP consensus statement recommends small bowel feeding if gastric residual volumes of 150ml or higher occur. The Canadian clinical practice guidelines recommend acceptance of gastric residual volumes up to 250 ml, use of prokinetic agents and jejunal feeding for patients, who are at high risk for intolerance of EN (on inotropes, sedatives, paralytic agents). When gastric enteral nutrition is insufficient despite acceptance of high gastric residual volumes and use of prokinetic agents, small bowel feeding is the best method to nevertheless feed the patient enterally because it is associated with a significant decrease of reflux, a reduced risk of aspiration and an adequate caloric intake.

For small bowel feeding the placement of a jejunal feeding tube is necessary. There are several possibilities to place the tube in the small bowel. An excellent method still is endoscopy, which has a success rate up to 98% and moreover allows an evaluation of the upper GI-tract concerning pathologies. However, it is a rather time consuming procedure, which is of limited availability and requires trained staff. As more simple alternatives unguided tubes and their placement in the small bowel were tested and showed success rates up to 75% only. One of these alternatives is a jejunal feeding tube, which is placed using an electromagnetic sensing technique to visualize the placement process on a bedside monitor (CORTRAK™). The aim of this study is the evaluation of the success rate of jejunal tube placement comparing the endoscopic versus the electromagnetic method in a comparative ICU patient population.

ELIGIBILITY:
Inclusion Criteria:

* Intolerance of intragastric feeding (high gastric residual volumes (≥250ml)and/or repeated vomiting)
* Clinical indication of jejunal feeding

Exclusion Criteria:

* Patients not fulfilling clinical indication of jejunal feeding or contraindications for jejunal feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Success rate of jejunal placement | 24h

SECONDARY OUTCOMES:
Time from initiation of tube placement till correct jejunal placement, time of tube in correct jejunal position, complications of placement | ICU-stay

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Department of Medicine III, ICU, Vienna, Austria

REFERENCES:
- [Derived] Holzinger U, Brunner R, Miehsler W, Herkner H, Kitzberger R, Fuhrmann V, Metnitz PG, Kamolz LP, Madl C. Jejunal tube placement in critically ill patients: A prospective, randomized trial comparing the endoscopic technique with the electromagnetically visualized method. Crit Care Med. 2011 Jan;39(1):73-7. doi: 10.1097/CCM.0b013e3181fb7b5f. PMID 21037470